CLINICAL TRIAL: NCT04267445
Title: A Prospective Single Centre Study to Evaluate the Safety and Effectiveness of Using Contrast Enhanced Ultrasound and Echogenic Embolic Agent Ekobi Embolization Microspheres in Prostate Artery Embolization for the Treatment of Men With Benign Prostatic Hypertrophy
Brief Title: Evaluate the Safety and Effectiveness of Using Echogenic Embolic Agent for Embolization of Prostate Artery for Treatment of Men With BPH (PAE CEUS)
Acronym: PAE CEUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: IMBiotechnologies Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: REB19-0963
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Embolization patients: Single center, open label, pilot study. Eligible patients will undergo transarterial embolization of the prostatic vasculature. Each patient will undergo a single embolization procedure.
  After completion of treatment in the first 2 patients and a review of follow-up assessments after 7 days, subsequent patients will be enrolled if no safety concerns have arisen in the first 2 patients.
  Ekobi Embolization MIcrospheres is administered via selective angiography and Prostatic Artery Embolization (PAE), a minimally invasive technique for reducing symptoms from Benign Prostatic Hyperplasia (BPH) to achieve near stasis in the target vasculature. Contrast Enhanced Ultrasound (CEU) and angiographic runs will be used to confirm anatomy at the time of embolization.
  Magnetic resonance imaging (MRI) and CEUS is used to assess changes in prostate volume and in central gland enhancement characteristics using 3D volume assessment software.
  Interventions: Procedure: Embolization of prostatic artery under ultrasound guidance

INTERVENTIONS:
Procedure: Embolization of prostatic artery under ultrasound guidance — Ekobi Embolization MIcrospheres is administered via selective angiography and Prostatic Artery Embolization (PAE), a minimally invasive technique for reducing symptoms from Benign Prostatic Hyperplasia (BPH) to achieve near stasis in the target vasculature. Contrast Enhanced Ultrasound (CEU) and angiographic runs will be used to confirm anatomy at the time of embolization.

SUMMARY:
A prospective single centre study to evaluate the safety and effectiveness of using contrast enhanced ultrasound and echogenic embolic agent Ekobi Embolization Microspheres in Prostate Artery Embolization for the Treatment of Men with Benign Prostatic Hyperplasia

DETAILED DESCRIPTION:
Single center, open label, pilot study. After screening and baseline testing, eligible patients will undergo transarterial embolization of the prostatic vasculature. Each patient will undergo a single embolization procedure.

After completion of treatment in the first 2 patients and a review of follow-up assessments after 7 days, subsequent patients will be enrolled if no safety concerns have arisen in the first 2 patients. Patients will be enrolled until 15 patients have undergone treatment. The patients will undergo MRI, contrast enhanced ultrasound and computerized tomography (CT) angiograpy/intra-procedural cone beam CT as required.

Ekobi Embolization MIcrospheres is administered via selective angiography and Prostatic Artery Embolization (PAE), a minimally invasive technique for reducing symptoms from Benign Prostatic Hyperplasia (BPH) to achieve near stasis in the target vasculature. Contrast Enhanced Ultrasound (CEU) and angiographic runs will be used to confirm anatomy at the time of embolization.

Magnetic resonance imaging (MRI) and CEUS is used to assess changes in prostate volume and in central gland enhancement characteristics using 3D volume assessment software.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be identified in the Urology Clinic diagnosed with benign prostatic hypertrophy and fit the criteria -

  1. Have received a diagnosis of BPH with moderate to severe LUTS, as determined by IPSS
  2. Are greater than 50 years of age
  3. Have had a pelvic examination by a urologist within the previous 6 months
  4. Have been refractory to medical therapy for 6 months, or have refused medical therapy
  5. Have a Qmax below 15 mL/s or acute urinary retention
  6. Prostate larger than 40 cm3
  7. Willing and able to provide written informed consent.

Exclusion Criteria:

* Patients will be excluded from this study if they meet any of the following criteria:

  1. Total serum PSA > 10.0 ng/mL at screening
  2. Advanced atherosclerosis and tortuosity of the iliac arteries
  3. PVR > 250 mL
  4. Use of phytotherapy for BPH within 2 weeks of screening visit
  5. Secondary renal insufficiency (due to prostatic obstruction)
  6. Chronic renal failure (glomerular filtration rate < 60)
  7. Large bladder diverticula or bladder stones
  8. Have claustrophobia or other contraindications to the performance of the pre- and post-procedure MRI studies, including but not confined to the presence of metal implants, metal plates, bone pins, bone screws, neurostimulators, cardiac pacemakers, aneurysm clips, cochlear or retinal implants, or permanent hearing aids
  9. Have compromised hematopoietic function (hemoglobin < 100 g/L; lymphocyte count < 500 x106/L; neutrophil count < 1.5 x 109/L; platelet count < 50 x 109/L
  10. Have had a documented anaphylactic reaction to a drug or anesthetic, or an allergic reaction to iodine contrast media not controlled by antihistamines or steroids
  11. Have received other investigational drugs or who have had experimental therapy within the past 4 weeks or are participating in any other concurrent experimental therapy
  12. Have abnormal coagulation profiles
  13. Are allergic to bovine collagen
  14. Are allergic to Perflutren 15 Are unable to comply with the follow up requirements of the study 16 Have serious cardiopulmonary compromise

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men have benign prostatic hyperplasia
Study Population: Men over 50 who have been diagnosed with benign prostatic hyperplasia and their prostates are larger than 40 cm3.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Dimensions of prostate | One year
  Measuring the prostate size in cm post treatment with embolization using the ultrasound guided embolization technique
Symptoms of benign prostate hyperplasia | One year
  Evaluate the efficacy of using contrast enhanced ultrasound and echogenic embolization agent Ekobi Embolization Microspheres on International Prostate Symptom Score (IPSS).

IPD SHARING:
Plan to Share IPD: No